CLINICAL TRIAL: NCT04532190
Title: Finding Alternatives to Standard Treatment for Attention-Deficit Hyperactivity Disorder
Acronym: FAST-ADHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Kara Murias, Assistant Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB20-1415
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
Keywords: Attention-Deficit/Hyperactivity Disorder (ADHD; Repetitive transcranial magnetic stimulation (rTMS)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active rTMS (Experimental): Active repetitive TMS
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Repetitive transcranial magnetic stimulation (rTMS)

SUMMARY:
Attention-Deficit/Hyperactivity Disorder (ADHD) is characterized by poor attention, impulsivity, hyperactivity and emotional-motivational dysregulation. Here, we will test if theta burst repetitive transcranial magnetic stimulation (rTMS) can reduce the symptoms of ADHD.

DETAILED DESCRIPTION:
Background & Rationale Attention-Deficit/Hyperactivity Disorder (ADHD) is characterized by poor attention, impulsivity, hyperactivity and emotional-motivational dysregulation. It has an estimated prevalence of 5% in children. Usually, ADHD in children is treated with stimulant medications, such as methylphenidate. However, these pharmacotherapy treatments have numerous unwanted side effects, including sleep disturbances, appetite changes, and emotional lability, and do not prove to be effective in every case.

A promising and alternative option for reducing ADHD symptoms is non-invasive brain stimulation. Repetitive transcranial magnetic stimulation (rTMS) is a form of non-invasive brain stimulation which involves the application of a magnetic field to the skull to change the behaviour and function of underlying brain areas. In turn, rTMS leads to positive long-term changes in neurochemical activity, and while studies are limited, some have shown that rTMS can reduce ADHD symptoms in adolescents with ADHD.

Methods Design: Open label TMS trial Primary Outcome: To examine the effect of active rTMS to the right prefrontal cortex on attention as measured by the TEACh-2

Outline:

1. Baseline Assessment (MRI Scan, assessment scales, neuropsychological testing)
2. rTMS intervention: 5 / week for 4 weeks.
3. Post-intervention Assessment (MRI Scan, assessment scales, neuropsychological testing).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ADHD
2. 9-15 years old
3. IQ greater than 80
4. English fluency (to enable consent/assent)
5. If on medication, must have been on the same type and dosage for at least 3 months.

Exclusion Criteria:

1. Diagnosis of mania, psychosis, or bipolar disorder
2. Impediments to TMS or MRI (i.e. metal implants in body)
3. Prior electroconvulsive therapy or vagus nerve stimulation
4. Diagnosis of Autism Spectrum Disorder.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
TEACH-2 | Baseline to week 5
  Test of everyday attention in children - 2. Direct assessment of attention abilities in children.

SECONDARY OUTCOMES:
SNAP-18 | 5 weeks and 52 weeks.
  Parent reporting of ADHD symptom severity
PedsQL | Baseline to week 5
  Self reporting of quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
If we do make individual participant data (IPD) available to other researchers it will be in keeping with local provincial laws on health information privacy. Data (if available) will be provided upon request.